CLINICAL TRIAL: NCT05499455
Title: Positional Therapy for the Treatment of Positional Obstructive Sleep Apnea in Children
Brief Title: SleepPOSAtive Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Indra Narang, Senior Associate Scientist, The Hospital for Sick Children
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: REB1000077578
Record Dates: First submitted 2022-08-10; First posted 2022-08-12 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Obstructive Sleep Apnea of Child

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Active Control
  Interventions: Device: Control
- Positional Sleep Belt (Experimental): Rematee Positional Sleep Belt
  Interventions: Device: Positional Sleep Belt

INTERVENTIONS:
Device: Positional Sleep Belt — Rematee Positional Sleep Belt
  Arms: Positional Sleep Belt
Device: Control — Control Device
  Arms: Control

SUMMARY:
This is a randomized crossover trial of children diagnosed with positional obstructive sleep apnea (POSA) on a baseline polysomnogram (PSG). Participants will undergo two further PSGs in random order over 4 weeks to assess the efficacy of a positional sleep therapy belt compared to a control for treating POSA.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is highly prevalent, and the gold standard therapy is continuous positive airway pressure (CPAP) for persistent OSA. Although CPAP is highly efficacious, long-term effectiveness is limited by poor adherence rates. Given the burden of untreated OSA in children, novel alternative therapies that are effective, acceptable and comfortable are urgently required.

OSA is characterized by recurrent obstruction of the upper airway associated with intermittent hypoxia and chronic sleep deprivation. OSA occurs in 1-4% of healthy children and in up to 80% of children with medical complexity (e.g. Down syndrome). It has significant health, societal, and economic impacts. CPAP is the gold standard therapy for persistent OSA but is poorly tolerated.

There is distinct clinical phenotype of OSA characterized by the predominance of obstructions in supine position, as measured by the obstructive apnea-hypopnea index (OAHI) on polysomnography (PSG). Up to half of children with OSA meet criteria for this phenotype which is termed positional OSA. Positional sleep belts that prevent children from adopting supine position may be beneficial for treating OSA but have not yet been studied in children.

The primary aim of this study is to assess the efficacy of a body positional sleep belt for the treatment of moderate to severe positional OSA in a paediatric population. This is a randomized crossover trial of children aged 4-18 years diagnosed with positional OSA. Participants will undergo two PSGs in random order over 4 weeks with a control and positional device therapy to assess treatment efficacy. Perceived comfort will be evaluated with surveys.

This novel research addresses a critical knowledge gap regarding the rigorous evaluation of alternative therapies beyond CPAP for managing OSA. Positional therapy has the potential to change clinical practice as an effective, cost-efficient, and non-invasive treatment option for children with positional OSA, particularly for children intolerant of CPAP.

ELIGIBILITY:
Inclusion Criteria:

1. Consent provided by patient or caregiver. If consent provided by caregiver, assent will be provided from patient whenever possible.
2. Children aged 4 to 18 years old
3. A diagnostic polysomnogram with obstructive apnea-hypopnea index of 5-30 events/hour.
4. Diagnosed with positional obstructive sleep apnea on baseline diagnostic polysomnogram as defined as:

   1. supine-to-nonsupine obstructive apnea-hypopnea index ratio of 2 or greater
   2. 10-90% total sleep time in supine position

Exclusion Criteria:

1. Current upper respiratory tract infection
2. Requires bilevel positive airway pressure in the opinion of the child's physician (e.g. diagnosed with co-existing central sleep apnea, chronic respiratory failure, or bradypnea for age)
3. Requiring oxygen therapy
4. Unable to reposition independently
5. Total sleep time < 4 hours on diagnostic polysomnogram
6. Unable to tolerate electroencephalogram montage on diagnostic polysomnogram
7. Adherent to continuous positive airway pressure therapy (> 6 hours nightly usage)
8. Distance travelled to study site > 200 km

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2022-02-13 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2023-04-25 (Actual)

PRIMARY OUTCOMES:
Obstructive apnea-hypopnea index | 3 months
  Difference in obstructive apnea-hypopnea index with positional therapy versus control

SECONDARY OUTCOMES:
Comfort score | 3 months
  Difference in comfort score with positional therapy versus control. This is measured on a numeric rating scale with a score range of 0-10, with higher scores indicating decreased comfort.
Arousal index | 3 months
  Difference in arousal index with positional therapy versus control
Oxygen desaturation index | 3 months
  Difference in oxygen desaturation index with positional therapy versus control
Percentage of total sleep time supine | 3 months
  Difference in percentage of total sleep time supine with positional therapy versus control

CONTACTS AND LOCATIONS:
Overall Officials: Indra Narang, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xiao L, Baker A, Massicotte C, Reyna ME, Shi J, Wolter NE, Propst EJ, Mahant S, Amin R, Parekh RS, Narang I. Positional therapy for the treatment of positional obstructive sleep apnea in children: A randomized controlled crossover trial. Sleep Med. 2025 Jun;130:48-55. doi: 10.1016/j.sleep.2025.03.022. Epub 2025 Mar 28. PMID 40174291